CLINICAL TRIAL: NCT05897515
Title: LIAISON NES Flu A/B & COVID-19 Clinical Agreement in Australia
Brief Title: LIAISON NES Influenza (FLU) A/B & Coronavirus Disease 2019 (COVID-19) Clinical Agreement in Australia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DiaSorin Molecular LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DSM-PROT-005131
Record Dates: First submitted 2023-06-07; First posted 2023-06-09 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Influenza A; Influenza Type B; Coronavirus Disease 2019
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Masking Description: Participants are not provided investigational results and will only be provided with routine standard of care diagnostics results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blinded, Prospective Arm (Other): Clinical specimens shall be collected prospectively from patients with signs or symptoms of respiratory tract infection. Nasal swab in Copan universal transport media (UTM) 3 milliliters for comparator testing should be collected by a healthcare professional.
  Where subjects are willing and able, up to 40% of nasal swab for the investigational device will be self-collected under the guidance and supervision of a healthcare professional.
  Nasopharyngeal (NPS) specimens (optional) should only be collected by a healthcare professional. All specimens collected from children 13 years or younger should only be collected by a trained healthcare professional. Follow the Centers for Disease Control and Prevention guidelines for collecting NPS swabs, unless otherwise specified by the sponsor.
  Interventions: Diagnostic Test: LIAISON NES FLU A/B & COVID-19

INTERVENTIONS:
Diagnostic Test: LIAISON NES FLU A/B & COVID-19 — The LIAISON® NES FLU A/B & COVID-19 assay used on the LIAISON® NES instrument is a real-time PCR system that enables the direct amplification, detection and differentiation of Flu A viral RNA, Flu B viral RNA and SARS-CoV-2 RNA from dry nasal swabs. Nasal Swabs can be professionally collected by a Healthcare Provider or self-collected by the patient under the supervision of the healthcare provider. The collected nasal swab can then be directly loaded into the cartridge without nucleic acid extraction.

SUMMARY:
The DiaSorin Molecular LIAISON® NES FLU A/B & COVID-19 real-time polymerase chain reaction (RT-PCR) assay is intended for use on the DiaSorin LIAISON® NES instrument for the in-vitro qualitative detection and differentiation of nucleic acid from influenza A, influenza B and SARS-CoV-2 virus from dry nasal swabs (NS) from human patients with signs and symptoms during the acute phase of respiratory tract infection in conjunction with clinical and epidemiological risk factors.

The LIAISON® NES FLU A/B & COVID-19 assay is intended for use as an aid in the differential diagnosis of influenza A, influenza B and SARS-CoV-2 infection in a professional laboratory setting.

Negative results do not preclude influenza A, influenza B, or SARS-CoV-2, infection and should not be used as the sole basis for patient management decisions. The assay is not intended to detect the presence of the influenza C virus.

ELIGIBILITY:
Inclusion Criteria:

* Human patients with active signs and symptoms of respiratory tract infection at time of collection
* Specimens collected within 7 days of symptom onset for the initial collection
* Availability of age, gender, race, ethnicity, collection dates, collection time, routine respiratory testing method, routine respiratory result, signs and symptoms (e.g., fever), date of symptom onset for each symptom, vaccination status (Flu and COVID-19, as applicable), pre-existing medical conditions (as applicable), medications (e.g., COVID-19 antivirals), etc. for each subject

Exclusion Criteria:

* Incorrect swab type
* Incorrect transport media
* Incorrect specimen handling (specimens not stored at recommended temperature)
* Samples collected >7 days from symptom onset
* Subjects not consented

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | Samples will be tested on LIAISON NES within one hour of collection.
  Estimates of Sensitivity/percent positive agreement (PPA) and Specificity/percent negative agreement (NPA) will be calculated based on a two-by-two table (comparator method result vs. result from LIAISON® NES FLU A/B, RSV & COVID-19 assay or LIAISON PLEX® RSP Flex assay) for each target. In addition, 95% two-sided confidence intervals will be provided. A separate Sensitivity/PPA and Specificity/NPA for each target, to include those specimens excluded due to a discrepancy between the standard-of-care and molecular comparator result, will be presented in a separate 2 x 2 table.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Farhang, PhD, Principal Investigator — DiaSorin Molecular/Luminex Corporation
Locations (1):
- Grampians Health, Ballarat, Victoria, Australia